CLINICAL TRIAL: NCT05834738
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study of Atrasentan in Subjects With IgA Nephropathy on Sodium-glucose Cotransporter-2 Inhibitors (SGLT2i)
Brief Title: Randomized, Double-blind, Placebo-controlled, Crossover Study of Atrasentan in Subjects With IgA Nephropathy
Acronym: ASSIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CEXV811A12201; CHK01-03 (Other: Chinook Therapeutics Inc.); NCT06841094 (obsolete NCT alias)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy; Immunoglobulin A Nephropathy
Keywords: Kidney Diseases; Kidney Disease, Chronic; Urologic Diseases; Glomerulonephritis; Glomerular Disease; Glomerulonephritis, IGA; Glomerulopathy; Immunoglobulin Disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Renal Insufficiency, Chronic; Urologic Diseases; Glomerulonephritis | interventions — Atrasentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): Once daily oral administration of 0.75 mg atrasentan for 12 weeks (Period A) followed by once daily oral administration of placebo for 24 weeks (Period B)
  Interventions: Drug: Atrasentan; Drug: Placebo
- Sequence BA (Experimental): Once daily oral administration of placebo for 12 weeks (Period B) followed by once daily oral administration of 0.75 mg atrasentan for 24 weeks (Period A)
  Interventions: Drug: Atrasentan; Drug: Placebo

INTERVENTIONS:
Drug: Atrasentan — Period A (12 Weeks) - Film-coated tablet, Washout Period: 12 weeks, Period B (24 Weeks) - Placebo
  Other Names: CHK-01; Atrasentan Hydrochloride; ABT-627
  Arms: Sequence AB
Drug: Atrasentan — Period B (12 Weeks) - Placebo, Washout Period: 12 weeks, Period A (24 Weeks) - Film-coated tablet
  Other Names: CHK-01; Atrasentan Hydrochloride; ABT-627
  Arms: Sequence BA
Drug: Placebo — Placebo

SUMMARY:
The ASSIST study is a phase 2, double-blind, placebo-controlled crossover study to evaluate the safety and efficacy of atrasentan vs. placebo in subjects with IgA nephropathy (IgAN) while on background standard of care therapy and an SGLT2 inhibitor (SGLT2i).

DETAILED DESCRIPTION:
Approximately 52 patients with biopsy-proven IgAN who are on a background SGLT2i and a maximally tolerated and stable dose of a renin-angiotensin system inhibitor (RASi) [such as angiotensin converting enzyme inhibitor (ACEi) or angiotensin-receptor antagonist (ARB)] as part of standard of care, will be randomized to either sequence AB or sequence BA in which they will receive 0.75 mg atrasentan once daily during one period (period A), complete a 12-week washout period, and then receive matching placebo during the other period (period B) as determined by the randomization schema.

Subjects who are not on background SGLT2i therapy must be willing to undergo a run-in period of 8 weeks with an SGLT2i with a 24-hour total urine protein of > 0.85 grams/day at screening prior to the run-in period and have 24-hour total urine protein of > 0.5 grams/day at the end of the run-in period to be eligible for randomization.

Subjects will remain on their maximally tolerated and stable dose of RASi and stable dose of SGLT2i therapies for the duration of the study following randomization.

The primary objective of the study is to evaluate the efficacy of atrasentan vs. placebo while on background therapy with SGLT2i.

Subjects will have safety and efficacy assessments for 1 year (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Legal adults (per local and country specifications) ≥ 18 years of age at the time of signing the informed consent form (ICF) prior to initiation of any study specific activities/procedures.
* Biopsy-proven IgA nephropathy.
* Receiving a maximally tolerated and stable dose of a RASi for at least 12 weeks prior to screening. Investigator discretion should be used in determining maximally tolerated and optimized dose.
* eGFR of at least 30 mL/min/1.73 m^2 at screening based on the 2021 CKD-EPI equation.
* Willing to agree to highly effective forms of contraception, as specified in the protocol, throughout the study and for up to 1 month afterward. In WOCBP, use of hormonal contraceptive agents must have been started at least 1 month prior to baseline.
* Willing and able to provide informed consent and comply with all study requirements.
* Inclusion Criteria for SGLT2i stable subjects

  * Receiving a stable dose of an SGLT2i for at least 8 weeks prior to screening
  * Must have a 24-hour urine protein of >0.5 grams/day.
* Inclusion Criteria for Run-In Subjects

  * Must have a 24-hour total urine protein of >0.85 grams/day at screening
  * Willing to participate in an 8-week run-in period with an SGLT2i (per Investigator choice)
* Additional Inclusion Criteria for Run-in Subjects at the end of Run-In

  * Must have completed the 8-week run-in period on a stable and well tolerated dose of an SGLT2i
  * Must have a 24-hour total urine protein of >0.5 grams/day confirmed at the Run-in Week 8 visit.
  * Must have an eGFR of ≥ 30 mL/min/1.73 m^2 based on the CKD-EPI equation at their Run-in Week 8 visit.

Exclusion Criteria:

* Current diagnosis with another chronic kidney disease, including diabetic kidney disease.
* History of kidney transplantation or other organ transplantation.
* Use of systemic immunosuppressant medications, such as steroids, for more than 2 weeks in the past 3 months.
* Blood pressure above 150 mmHg systolic or 95 mmHg diastolic as evaluated by the Investigator.
* Known history of heart failure or prior hospital admissions for conditions relating to fluid overload that in the opinion of the Principal Investigator or Sponsor might confound the results of the study or pose additional risk to the participant by their participation in the study.
* Clinically significant history of liver disease as assessed by the Investigator.
* Hemoglobin below 9 g/dL as measured by the Investigator or prior history of blood transfusion for anemia within the past 3 months.
* Malignancy within the past 5 years. Exceptions to this criteria include nonmelanoma skin cancer and curatively treated cervical carcinoma in situ.
* For women, pregnancy, breast feeding, or intent to become pregnant during the study. and at least 1 month afterward.
* For men, intent to father a child or donate sperm during the study.
* Have received any investigational agent or approved treatment for IgAN (other than a RAS inhibitor) including SGLT2i (except for subjects in the SGLT2i stable stratum) within 1 month (or 5 half-lives of the agent, whichever is longer) prior to Screening. If the investigational agent is a cytotoxic or immunosuppressive agent then this washout period is 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Proteinuria at Week 12 in Both Treatment Periods 1 and 2 | Baseline and 12 weeks or approximately 3 months
  The change in urine protein: creatinine ratio (UPCR) from baseline to Week 12

SECONDARY OUTCOMES:
Change From Baseline in Proteinuria at Week 24 in Treatment Periods 2 | Baseline and 24 weeks or approximately 6 months
  The change in UPCR from baseline to Week 24
Number of Subjects With Adverse Events (AEs) | From informed consent until end of study, approximately 60 weeks
  Type, incidence, severity, seriousness, and relatedness of AEs will be collected.
Plasma Concentration of Atrasentan | Treatment Period 1: Pre-dose on Weeks 2, 6 and 12; Treatment Period 2: Pre-dose on Weeks 2, 6, 12 and 24
  Blood samples will be collected for the measurement of plasma concentrations of atrasentan.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (6):
  - University of Alabama at Birmingham (UAB) - The Kirklin Clinic (TKC) - Nephrology Clinic, Birmingham, Alabama
  - Fides Clinical Research, Atlanta, Georgia
  - NANI Research, Oak Brook, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - University of North Carolina at Chapel Hill - Nephrology and Hypertension, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Australia (4):
  - The St. George Hospital, Kogarah, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Monash Health- Monash Medical Centre, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Brazil (4):
  - NUPEC Cardio, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Sao Paulo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo
- Malaysia (4):
  - Hopsital Sultanah Aminah Johor Bharu (HSAJB) - Bangunan Bakawali Heodialysis Centre, Johor Bahru, Johor Darul Takzim
  - Universiti Kebangsaan Malaysia (UKM) - Medical Centre (Pusat Perubatan) (Hospital Canselor Tuanku Muhriz (HCTM)), Cheras, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun (HRPB), Ipoh, Perak
- South Korea (4):
  - Dong-A University Medical Center (Dong-A University Hospital), Busan, Busan
  - Soon Chun Hyang Central Medical Center (SCHMC) - Soon Chun Hyang University Hospital, Cheonan, Chungnam-Do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Chung-Ang University College, Seoul, Seoul
- Spain (8):
  - Hospital Torrecardenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital del Vall d´Hebron, Barcelona
  - Hospital Ribera Polusa, Lugo
  - Hospital Universitario De Getafe (HUG), Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Virgen Macarena, Seville
  - Hospital Clinico Universitario, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639